CLINICAL TRIAL: NCT07329088
Title: ISOLeucine Addition Treatment Effects (ISOLATE) in a Controlled Diet Study
Brief Title: Isoleucine Addition Treatment Effects in a Controlled Diet Study
Acronym: ISOLATE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jean L. Fry (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor-Investigator, Jean L. Fry, Associate Professor-PI, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 108059; P20GM156679 (NIH)
Record Dates: First submitted 2026-01-07; First posted 2026-01-09 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-01

CONDITIONS: Prediabetes (Insulin Resistance, Impaired Glucose Tolerance); Metabolic Syndrome (MetS); Obesity & Overweight
Keywords: L-Isoleucine; Insulin Resistance; Hyperglycemia; Muscle, Skeletal; Amino Acids; Prediabetic State; Diet; Mechanistic Target of Rapamycin Complex 1; Adipose Tissue; Body Composition
MeSH Terms: conditions — Prediabetic State; Insulin Resistance; Glucose Intolerance; Metabolic Syndrome; Obesity; Overweight; Hyperglycemia | interventions — Isoleucine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Isoleucine group (Experimental): Participants will be randomized to receive low-isoleucine diet and isoleucine supplement
  Interventions: Dietary Supplement: L-Isoleucine; Other: Low-isoleucine diet
- Placebo group (Active Comparator): Participants will be randomized to receive low-isoleucine diet and placebo supplement
  Interventions: Other: Low-isoleucine diet

INTERVENTIONS:
Dietary Supplement: L-Isoleucine — Participants will follow a habitual American style diet. All participants transition to a healthy, low-isoleucine diet the study team provides, but only the isoleucine group receives isoleucine supplements to replete the overall diet to typical intake levels.
  Arms: Isoleucine group
Other: Low-isoleucine diet — Healthy, weight-maintaining, low-isoleucine meals and snacks will be provided directly to participants for 4 weeks. Diets are formulated by registered dietitians to meet energy, protein, and amino-acid requirements while minimizing weight change; target macronutrient distribution ≈ 10% protein / 60% carbohydrate / 30% fat38. Isoleucine content will meet minimum needs of 23 mg/kg.

SUMMARY:
The primary purpose of this study is to determine whether isoleucine repletion attenuates increases in insulin sensitivity typically observed when people with obesity follow a healthy, low-isoleucine diet.

DETAILED DESCRIPTION:
Isoleucine restriction promotes insulin sensitivity in preclinical models and is a promising strategy for preventing type 2 diabetes. This project aims to identify clinical and molecular changes in skeletal muscle and adipose tissues when adults with obesity switch from a typical American style diet to a plant-based diet low in isoleucine with or without isoleucine repletion.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥ 30
* Meeting at least three metabolic syndrome criteria
* Follow an American style diet

Exclusion Criteria:

* Type 1 or 2 Diabetes diagnosis
* Medical condition or medication that affects insulin sensitivity, weight, or metabolism
* More than 5% weight change in 3 previous months
* Restrictive dietary pattern
* History of bariatric surgery
* Food allergy more severe than grade 1 on the CoFAR Grading Scale for Systemic Allergic Reactions, Version 3.0
* Allergy to lidocaine.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-03-02 (Estimated); Primary Completion 2029-01-31 (Estimated); Study Completion 2029-01-31 (Estimated)

PRIMARY OUTCOMES:
Change in insulin sensitivity (M value) | The first measure is taken immediately after the run-in and the final measure will be taken immediately after the completion of the low-isoleucine diet and isoleucine vs placebo supplement intervention four weeks later.
  The primary clinical outcome is insulin sensitivity, quantified as the M value derived from the hyperinsulinemic-euglycemic clamp. Hyperinsulinemic-euglycemic clamps will be performed to measure insulin sensitivity (IS). Briefly, after a ≥8 hour fast, participants will be admitted to the PC clinical unit and two IVs will be inserted; one for infusion, the other for blood draws. The primary metric will be an absolute change in M value from baseline to post intervention.

SECONDARY OUTCOMES:
Change in ratio of phosphorylation IRS-1 in skeletal muscle | The first measure is taken immediately after the run-in and the final measure will be taken immediately after the completion of the low-isoleucine diet and isoleucine vs placebo supplement intervention four weeks later.
  Phosphorylation of IRS-1 at Ser636/639 will be quantified in skeletal muscle tissue obtained at baseline and after the intervention. Levels of phosphorylated IRS-1 and total IRS-1 will be measured, and the outcome will be expressed as the change in the phospho-to-total IRS-1 protein ratio from baseline to post-intervention.
Absolute change in visceral fat | The first measure is taken immediately after the run-in and the final measure will be taken immediately after the completion of the low-isoleucine diet and isoleucine vs placebo supplement intervention four weeks later.
  Abdominal adiposity will be assessed by computed tomography (CT). A single slice at the L4/L5level will be obtained at baseline and post-intervention. Visceral and subcutaneous fat volumes will be quantified using ImageJ.
Change in ratio of phosphorylation Akt in skeletal muscle | The first measure is taken immediately after the run-in and the final measure will be taken immediately after the completion of the low-isoleucine diet and isoleucine vs placebo supplement intervention four weeks later.
  Phosphorylation of Akt (Thr308 and Ser473) will be quantified in skeletal muscle tissue obtained at baseline and after the intervention. Levels of phosphorylated Akt and total Akt will be measured, and the outcome will be expressed as the change in the phospho-to-total Akt protein ratio from baseline to post-intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Jean Fry, PhD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Doi M, Yamaoka I, Fukunaga T, Nakayama M. Isoleucine, a potent plasma glucose-lowering amino acid, stimulates glucose uptake in C2C12 myotubes. Biochem Biophys Res Commun. 2003 Dec 26;312(4):1111-7. doi: 10.1016/j.bbrc.2003.11.039. PMID 14651987
- [Background] Zhang S, Yang Q, Ren M, Qiao S, He P, Li D, Zeng X. Effects of isoleucine on glucose uptake through the enhancement of muscular membrane concentrations of GLUT1 and GLUT4 and intestinal membrane concentrations of Na+/glucose co-transporter 1 (SGLT-1) and GLUT2. Br J Nutr. 2016 Aug;116(4):593-602. doi: 10.1017/S0007114516002439. PMID 27464458
- [Background] Woo SL, Yang J, Hsu M, Yang A, Zhang L, Lee RP, Gilbuena I, Thames G, Huang J, Rasmussen A, Carpenter CL, Henning SM, Heber D, Wang Y, Li Z. Effects of branched-chain amino acids on glucose metabolism in obese, prediabetic men and women: a randomized, crossover study. Am J Clin Nutr. 2019 Jun 1;109(6):1569-1577. doi: 10.1093/ajcn/nqz024. PMID 31005973
- [Background] Drummond MJ, Bell JA, Fujita S, Dreyer HC, Glynn EL, Volpi E, Rasmussen BB. Amino acids are necessary for the insulin-induced activation of mTOR/S6K1 signaling and protein synthesis in healthy and insulin resistant human skeletal muscle. Clin Nutr. 2008 Jun;27(3):447-56. doi: 10.1016/j.clnu.2008.01.012. Epub 2008 Mar 14. PMID 18342407
- [Background] Yu D, Richardson NE, Green CL, Spicer AB, Murphy ME, Flores V, Jang C, Kasza I, Nikodemova M, Wakai MH, Tomasiewicz JL, Yang SE, Miller BR, Pak HH, Brinkman JA, Rojas JM, Quinn WJ 3rd, Cheng EP, Konon EN, Haider LR, Finke M, Sonsalla M, Alexander CM, Rabinowitz JD, Baur JA, Malecki KC, Lamming DW. The adverse metabolic effects of branched-chain amino acids are mediated by isoleucine and valine. Cell Metab. 2021 May 4;33(5):905-922.e6. doi: 10.1016/j.cmet.2021.03.025. Epub 2021 Apr 21. PMID 33887198
- [Background] Yeh CY, Chini LCS, Davidson JW, Garcia GG, Gallagher MS, Freichels IT, Calubag MF, Rodgers AC, Green CL, Babygirija R, Sonsalla MM, Pak HH, Trautman M, Hacker TA, Miller RA, Simcox J, Lamming DW. Late-life isoleucine restriction promotes physiological and molecular signatures of healthy aging. bioRxiv [Preprint]. 2024 Jan 9:2023.02.06.527311. doi: 10.1101/2023.02.06.527311. PMID 36798157
- [Background] Trautman ME, Richardson NE, Lamming DW. Protein restriction and branched-chain amino acid restriction promote geroprotective shifts in metabolism. Aging Cell. 2022 Jun;21(6):e13626. doi: 10.1111/acel.13626. Epub 2022 May 8. PMID 35526271
- [Background] Green CL, Trautman ME, Chaiyakul K, Jain R, Alam YH, Babygirija R, Pak HH, Sonsalla MM, Calubag MF, Yeh CY, Bleicher A, Novak G, Liu TT, Newman S, Ricke WA, Matkowskyj KA, Ong IM, Jang C, Simcox J, Lamming DW. Dietary restriction of isoleucine increases healthspan and lifespan of genetically heterogeneous mice. Cell Metab. 2023 Nov 7;35(11):1976-1995.e6. doi: 10.1016/j.cmet.2023.10.005. PMID 37939658
- [Background] Fontana L, Cummings NE, Arriola Apelo SI, Neuman JC, Kasza I, Schmidt BA, Cava E, Spelta F, Tosti V, Syed FA, Baar EL, Veronese N, Cottrell SE, Fenske RJ, Bertozzi B, Brar HK, Pietka T, Bullock AD, Figenshau RS, Andriole GL, Merrins MJ, Alexander CM, Kimple ME, Lamming DW. Decreased Consumption of Branched-Chain Amino Acids Improves Metabolic Health. Cell Rep. 2016 Jul 12;16(2):520-530. doi: 10.1016/j.celrep.2016.05.092. Epub 2016 Jun 23. PMID 27346343